CLINICAL TRIAL: NCT03100643
Title: Development of a Couple-Based Mobile Health Intervention for Enhancing HIV Care Engagement Outcomes (N'Gage)
Acronym: N'Gage
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 5K01MH106416-02 (NIH)
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS, mHealth, intervention development, African American men
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: mHealth N'Gage mobile application — To enhance HIV care engagement among couples using mobile technology.

SUMMARY:
HIV/AIDS among Black men is a US public health crisis, emphasizing the urgency for increased research focus and intervention development. The overall objective of this application is to achieve a better understanding of the role that dyadic factors play in individual-level HIV care engagement outcomes among HIV-positive Black men in romantic relationships. The end goal is the development of an intervention that employs innovative mobile technology to target partnership dynamics that optimize outcomes in the HIV care continuum.

DETAILED DESCRIPTION:
Compared to other racial/ethnic groups in the US, Black men who have sex with men (MSM), once diagnosed, are less likely to be optimally engaged in HIV care and treatment. This undermines the promise of prevention approaches for reducing the disproportionate effects of HIV/AIDS on Black communities, emphasizing the urgency for increased research focus and intervention development. Understanding HIV care engagement in the context of the dyad may be part of a comprehensive effort to addressing multilevel influences on HIV care engagement that are unique to HIV+ Black MSM towards achieving the maximum public health benefit of treatment-as-prevention. However, the scarcity of dyad-level research limits our understanding of dyadic effects HIV care engagement to inform intervention development. Mobile technology-based strategies (mHealth) offer tremendous potential as an acceptable, feasible, and effective intervention approach for enhancing HIV care engagement among partnered HIV+ Black MSM for several important reasons: (1) Black MSM are likely to report having a primary partner and to participate in couple-based HIV interventions; (2) couple-based behavior (e.g., daily routines of the couple), within-partnership dynamics (e.g., trust, intimacy), and couple serostatus (i.e., serodiscordant and concordant-positive relationships) are understudied factors in optimal HIV care engagement among MSM; and (3) mHealth has shown feasibility and acceptability in targeting couple-based behavior (e.g., money management, family planning) in the general population. Moreover, mHealth offers potential in addressing social and structural barriers often experienced by Black MSM in accessing and engaging in HIV care. Therefore, the aims of the study are to: (Aim 1) examine mobile technology use and relational factors involved in HIV care engagement within the context of couples among HIV+ Black MSM; (Aim 2) synthesize Aim 1 findings to identify intervention targets for behavioral change and to derive a framework of an intervention to enhance HIV care engagement in a dyadic context; and (Aim 3) develop a novel, mobile technology product for enhancing HIV care engagement in the context of couples among HIV+ Black MSM. The end goal of the application is the development of a novel, theory-based, user-centered mHealth product that targets relationship factors and dynamics important in optimal HIV care engagement among HIV+ Black men in same-sex relationships. Through these aims, I will acquire additional training necessary for my career development in (a) theory and research methods (qualitative research methods and dyadic analysis) for conducting couple-based research, (b) formative research in intervention development using group model building, and (c) mHealth product development. These research and career development activities will build the foundation to my becoming an independent, NIH-funded investigator with skills to conduct couple-based intervention research using mobile health innovations that is part of a comprehensive effort in HIV prevention integrating advances in mobile technology and behavioral medicine to reduce racial/ethnic disparities in HIV.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as African American or Black
* Identifies with and presents as male
* Is currently in a committed romantic relationship
* Is HIV-positive
* Have access to a mobile phone that can access the Internet

Exclusion Criteria:

* None.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identify as male.
Study Population: HIV-positive African American sexual minority men in a primary relationship and their relationship partner.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Qualitative interview data on how participants used and liked the mHealth intervention prototype. | Outcomes will be measured after a two-week pilot period during the fourth year of the project.
  Outcome will be based on qualitative feedback on prototype design, e.g., the look and feel of the prototype, how often the participants interacted with the prototype features, and whether or not participants feel that the intervention would be useful or helpful in improving their engagement in HIV care.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States